CLINICAL TRIAL: NCT00885014
Title: Telephone Cognitive-behavioral Therapy for Subthreshold Depression and Presenteeism in Workplace: a Randomized Controlled Trial
Brief Title: Telephone Cognitive-Behavioral Therapy (CBT) for Subthreshold Depression and Presenteeism in Workplace
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyoto University (Other)
Collaborators: Nagoya City University (Other)
Responsible Party: Principal Investigator, Toshiaki A. Furukawa, Professor, Kyoto University
Organization: Kyoto University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCUPsychiatry002
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: Depressive disorder; Behavior therapy; Workplace; Subthreshold depression
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT (Experimental): Telephone cognitive-behavioral therapy
  Interventions: Behavioral: CBT; Behavioral: EAP
- TAU (Active Comparator): Treatment as usual through the Employees Assistance Program
  Interventions: Behavioral: EAP

INTERVENTIONS:
Behavioral: CBT — Telephone cognitive-behavioral therapy
  Arms: CBT
Behavioral: EAP — Employees Assistance Program

SUMMARY:
The purpose of the study is to examine the effectiveness of telephone cognitive-behavioral therapy for subthreshold depression and presenteeism in workplace, in comparison with treatment-as-usual (TAU) (which is minimal contact through Employers Assistance Program (EAP)).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-57 at study entry [because the retirement age is usually 60, we have to recruit the patients well before 60 in order to allow time for follow-up]
* Men and women
* Currently employed full-time (either regular or temporary) by the business company
* Expected to be employed full-time for 2 years after screening
* K6 scores greater than or equal to 9 (or 10) at screening
* BDI2 scores greater than or equal to 10 at 2nd screening (Composite International Diagnostic Interview (CIDI) interview)

Exclusion Criteria:

* Part-time employees
* Sick leave for 6 or more days for a physical or mental condition in the past month
* Expected to be on pregnancy leave, maternity leave or nursing leave within 2 years after screening
* Current treatment for a mental health problem from a mental health professional
* Major depressive episode in the past month, as ascertained by CIDI [We do not exclude dysthymia or major depression in partial remission]
* Lifetime history of bipolar disorder, as ascertained by CIDI
* Any substance dependence in the past 12 months, as ascertained by CIDI. [We do not exclude substance abuse.]
* Any other current mental disorder if it constitutes the predominant aspect of the clinical presentation and requires treatment not offered in the project
* Those who have already received the telephone CBT in the pilot runs

Ages: 20 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Depression severity as measured by Beck Depression Inventory-II (BDI2) | 4 months post-randomization
Work performance as measured by the Health and Work Performance Questionnaire (HPQ) "effective hours worked" for the past month | 4 months post-randomization

SECONDARY OUTCOMES:
Depression severity as measured by Kessler Scale (K6) | 4 months post-randomization
Client satisfaction as measured by Visual Analogue Scale (VAS) | 4 months post-randomization
Depression severity as measured by BDI2 and K6 | 15 months post-randomization
Work performance as measured by HPQ and by job retention | 15 months post-randomization
Client satisfaction as measured by VAS | 15 months post-randomization
Use of EAP services and other health services | 15 months post-randomization
Suicidal attempt and/or hospitalization (physical or mental) | 15 months post-randomization
Time to incident major or minor depressive episode | 15 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Furukawa, MD, PhD, Principal Investigator — Nagoya City University
Locations (1):
- Nagoya City University, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Hayasaka Y, Furukawa TA, Sozu T, Imai H, Kawakami N, Horikoshi M; GENKI Project. Enthusiasm for homework and improvement of psychological distress in subthreshold depression during behavior therapy: secondary analysis of data from a randomized controlled trial. BMC Psychiatry. 2015 Nov 25;15:302. doi: 10.1186/s12888-015-0687-3. PMID 26602093
- [Derived] Furukawa TA, Horikoshi M, Kawakami N, Kadota M, Sasaki M, Sekiya Y, Hosogoshi H, Kashimura M, Asano K, Terashima H, Iwasa K, Nagasaku M, Grothaus LC; GENKI Project. Telephone cognitive-behavioral therapy for subthreshold depression and presenteeism in workplace: a randomized controlled trial. PLoS One. 2012;7(4):e35330. doi: 10.1371/journal.pone.0035330. Epub 2012 Apr 19. PMID 22532849